CLINICAL TRIAL: NCT05909917
Title: Deploying Emergency Bystander Internet Training (DEBIT) for Lay First Responders in Resource Limited Settings
Brief Title: Deploying Emergency Bystander Internet Training
Acronym: DEBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: LFR International (Unknown)
Responsible Party: Principal Investigator, Zachary Eisner, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00228774
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Trauma; Trauma Injury
Keywords: Pre-Hospital; First Responder; First Aid; Education
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to intervention arm randomization of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person (Active Comparator): Participants will undergo a previously validated, half-day first responder training course, taught live in-person by local instructors in each study location. Participant knowledge acquisition will be measured via a 23-question pre/post-training assessment, administered in person. Participant skill performance will be measured via direct observation grading of a standardized patient encounter, performed in person.
  Interventions: Other: Half-Day First Responder Training
- Virtual (Experimental): In a controlled computer laboratory setting, participants will undergo an experimental first responder training course consisting of a half-day of pre-recorded video, lecture notes, and illustrations. Participant knowledge acquisition will be measured via a 23-question pre/post-training assessment, administered in person. Participant skill performance will be measured via direct observation grading of a standardized patient encounter, performed in person.
  Interventions: Other: Half-Day First Responder Training

INTERVENTIONS:
Other: Half-Day First Responder Training — Participants in both study arms will undergo a half-day first responder training course designed for laypeople. The course will consist of five curricular categories: scene management, airway and breathing, hemorrhage control, fracture management, and victim transport. Course material will not differ between in-person and virtual arms, however the method of information dissemination will vary.

SUMMARY:
The primary aim of this study is to evaluate the efficacy of a massive open online course (MOOC) for training lay first responders in sub-Saharan Africa. The research team will assess educational outcomes of first responder training implemented at program locations in Nigeria, Sierra Leone, Uganda, and Kenya, through previously validated pre- and post-course survey instruments, standardized patient assessments, and incident reporting. The research team will investigate efficacy of MOOC training amongst diverse populations with variable technology literacy and utilize data gathered to develop more efficient means of disseminating basic first aid training information.

DETAILED DESCRIPTION:
Low- and middle-income countries (LMIC) bear the brunt of non-intentional traumatic injury. In fact, millions of people die from injury each year, with 90% of the mortality faced by LMICs. An additional 650 million people suffer from disabilities resulting from similar causes worldwide. The expansion of emergency medical services (EMS) in low- and middle-income countries could address 45% of all deaths and 36% of the total disease burden in low-income countries. However, emergency care, let alone prehospital emergency medical services, are often not priorities in LMICs. Though injury is the leading prehospital condition in Africa, 91.3% of the African population has no EMS available and there is no evidence of EMS systems in 61% of African countries. Sub-Saharan Africa is particularly affected, as available data on emergency care demonstrates the current combination of high patient volume and mortality make emergency care an urgent area of focus for future mortality-reducing interventions, especially as 80% of injury deaths occur in the prehospital setting in low-resource settings compared with just 59% in developed settings. Several studies investigating programs training lay first responders to treat the previously unaddressed traumatic injury burden were undertaken beginning in the mid- to late-1990's.

Subsequent to those initial studies, the World Health Organization (WHO) recommended establishing lay first responder systems as the first step toward developing formal emergency medical services in 2004. However, global uptake of the guidelines has been limited, even as injury has become the leading cause of death for young people between ages 15 and 45. Most LMICs lack organized EMS systems, while ambulances have been used primarily for interfacility transport, rather than as emergency care vehicles. Since the 2004 WHO announcement, many programs have attempted to leverage pre-existing networks of first responders, such as commercial drivers, lay persons, and bystanders, who currently already provide a large proportion of prehospital transport and occasionally also provide first aid in LMICs. As such, EMS system development since has been incongruous and varied, though the lay first responders (LFR) Model has demonstrated program success across heterogeneous across regions. Despite the World Health Organization recommendation and studies completed subsequently, the first aid provided by laypeople to victims of trauma requires additional programs and studies investigating first responder training, program scalability, and clinical implications for trauma patients. To meet these needs, the primary objectives of this study are to evaluate the educational efficacy and clinical impact of a Massive Open Online Course (MOOC) for LFR training through international roll-out.

A randomized control trial design with two arms will be identically deployed in four settings: Sierra Leone (Makeni), Nigeria (Lagos), Uganda (Mukono), and Kenya (Kakamega). In the control arm, participants will be assigned to a previously validated half-day first responder course and assessed for knowledge acquisition and clinical skills performance. In the experimental arm, participants will be assigned to a novel half-day MOOC course and similarly assessed for knowledge acquisition and clinical skills performance. Trainees in both arms will be monitored for knowledge retention and skill usage post-training. Outcomes will demonstrate the relative efficacy of the novel MOOC course as compared to traditional in-person training methods, and may inform LFR program scalability in future EMS capacity building efforts.

ELIGIBILITY:
Inclusion Criteria:

- Commercial transportation providers

Exclusion Criteria:

- Does not possess means of transportation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Knowledge Acquisition | 3 months
  Acquisition will be measured using a 23-question test administered prior to the intervention and then immediately following training. Scores for the test range from 0 (no knowledge acquired) to 23 (all knowledge acquired).
Clinical Skills Performance Checklist - Airway Management | 3 months
  Performance will be assessed using a direct-observation checklist evaluating first-responder interventions on standardized patients. Participants will be assessed on one of two clinical scenarios: airway management and fracture management. The airway management checklist will have a total of 8 points with higher score indicating better performance (0-8, with 0 meaning failed performance and 8 meaning perfect performance).
Clinical Skills Performance Checklist - Fracture Management | 3 months
  Performance will be assessed using a direct-observation checklist evaluating first-responder interventions on standardized patients. Participants will be assessed on one of two clinical scenarios: airway management and fracture management. The fracture management checklist will have a total of 12 points with higher score indicating better performance (0-12, with 0 meaning failed performance and 12 meaning perfect performance).

SECONDARY OUTCOMES:
Knowledge Retention | 9 months
  Retention will be measured using the same 23-question test used to assess knowledge acquisition but administered at 6 months and then 9 months following the intervention. Scores for the test range from 0 (no retention) to 23 (all knowledge retained).
Skill Usage | 6 months
  Usage will be tracked using incident report forms where participants reported using the skills acquired from the intervention to treat someone. Incident report forms will include de-identified patient information, care rendered by the first responder, location of the treated injury, mechanism of the treated injury, injury severity, and the hospital transportation method employed.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Eisner, BS, Principal Investigator — University of Michigan
Locations (4):
- Masinde Muliro University of Science and Technology, Kakamega, Kakamega County, Kenya
- Health Emergency Initiative, Lagos, Lagos, Nigeria
- School of Clinical Sciences, Makeni, Northern Province, Sierra Leone
- Vision for Trauma Care in Africa, Mukono, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No